CLINICAL TRIAL: NCT04467918
Title: Cannabidiol (CBD) in Patients With Mild to Moderate Symptoms of Coronavirus 2019: A Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: CANnabiDiol for CoviD-19 pATiEnts With Mild to Moderate Symptoms
Acronym: CANDIDATE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Jose Alexandre de Souza Crippa, Professor of Psychiatry, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CANDIDATE study
Record Dates: First submitted 2020-07-03; First posted 2020-07-13 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: SARS-CoV2
Keywords: SARS-CoV2; Cannabidiol
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: A total of 104 patients with SARS-CoV-2 infection will be included in the study (i.e., 52 cases in the CBD group plus pharmacological and clinical measures and 52 in the placebo group plus pharmacological and clinical measures). All patients will receive the clinical and pharmacological measures standardized by the Brazilian Ministry of Health's practical guidelines for diagnosis and treatment for mild and moderate cases for SARS-CoV-2
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (CBD) (Experimental): 50 cases in the CBD group plus pharmacological and clinical measures. Patients in the investigational treatment group will receive CBD within 24 hours after randomization, with a daily dose of 300mg / day (two 150mg doses; 1mL of the formulation) for 14 days.
  Interventions: Drug: Cannabidiol
- Placebo (PLB) (Placebo Comparator): 50 in the placebo group plus pharmacological and clinical measures. Patients in the placebo group will also receive, within 24 hours after randomization, 1mL of the same investigational medication vehicle (medium / coconut chain triglyceride oil - MCT) for 14 days
  Interventions: Other: PLACEBO

INTERVENTIONS:
Drug: Cannabidiol — Already described
  Other Names: CBD
  Arms: Cannabidiol (CBD)
Other: PLACEBO — Already described
  Other Names: PLB
  Arms: Placebo (PLB)

SUMMARY:
The aim of this work is to conduct a randomized, double-blind, placebo-controlled clinical trial to assess the efficacy and safety of cannabidiol (CBD - 300 mg a day) in patients infected with SARS-CoV-2.

The specific objectives are to assess whether, in patients with mild and moderate forms of SARS-CoV-2, daily use of CBD 300 mg for fourteen days is capable of:

i) decrease viral load; ii) modify inflammatory parameters, such as cytokines, measured from serum; iii) reduce clinical and emotional symptoms through daily clinical evaluation; iv) improve sleep; v) reduce hospitalization and worsen the severity of the disease; v) Monitor the possible adverse effects of CBD use in these patients.

DETAILED DESCRIPTION:
The present study will be a single-center, randomized, parallel, double-blind, placebo-controlled clinical trial of CBD in patients with mild to moderate SARS-CoV-2 infection. The investigators will use random stratification by minimizing the sample to stratify all eligible patients according to gender, age, disease severity (mild or moderate) and presence of comorbidity (controlled diabetes and/or hypertension), followed by random designation (in a ratio 1: 1) in each stratum to ensure a balanced distribution of disease severity among treatment groups (CBD plus symptomatic clinical and pharmacological measures) and control (symptomatic clinical and pharmacological measures and placebo). All patients will receive the clinical and pharmacological measures standardized by the Brazilian Ministry of Health's practical guidelines for diagnosis and treatment for mild and moderate cases for SARS-CoV-2 (https://portalarquivos.saude.gov.br/images/pdf /2020/April/18/Dirursos-Covid19.pdf). In other words, the following pharmacological measures: "prescription of drugs for symptom control, if there is no contraindication, with the possibility of intercalating antipyretic drugs in cases of difficult control of fever. • Oral antipyretic: 1st option: Paracetamol 500-1000 mg/dose (maximum 3mg / day) • 2nd option: Dipyrone 500-1000 mg VO (maximum dose in adults 4 grams)", and clinical measures:" Home isolation by 14 days from the date of onset of symptoms; review every 48 hours, preferably by phone, providing face-to-face assistance, if necessary; maintain rest, a balanced diet and a good supply of fluids; isolation from home contacts for 14 days".

Thus, all patients will receive clinical and pharmacological measures of symptoms. Patients in the investigational treatment group will also receive CBD within 24 hours after randomization, with a daily dose of 300mg / day (two 150mg doses; 1mL of the formulation) for 14 days. Patients in the placebo group will also receive, within 24 hours after randomization, 1mL of the same investigational medication vehicle (medium/coconut chain triglyceride oil - MCT) for 14 days, using a dosing device/syringe indistinguishable from the CBD medication. Patients, nursing staff, laboratory technicians, doctors who will carry out the assessments, researchers, and statisticians will be blind to the treatment group and will not know about the treatment information.

Secretions from the upper respiratory tract, lower respiratory tract, or both, by swab, will be obtained from each patient in the screening (day -3 to day 1) during treatment and post-treatment follow-up at the patient's home on days 1, 2, 3, 4, 5, 7, 10, 14, 21, and 28, to test the viral load and SARS-CoV-2 genotyping. On all these dates, nurses will visit home to collect swab (only from the oropharynx, to minimize discomfort), blood and will be evaluated at each visit for vital signs, pulse oximetry, odor test, and treatment guidelines. Each patient will also receive a digital thermometer to measure the axillary temperature in case of suspected fever and daily measurement immediately before lunch and dinner.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes, older than 18 years of age, with SARS-CoV-2 infection confirmed in upper or lower respiratory tract secretion, through reverse transcription followed by polymerase chain reaction (RT- PCR), with mild or moderate manifestations of Covid-19, who wish to participate, and consent by signing the informed consent form and not involved in another clinical trial during the study period
2. Pneumonia assessed clinically and / or radiologically will not be mandatory for inclusion
3. Have a telephone (cellular or landline) that may be available to receive daily calls throughout the study period.
4. Willingness to voluntarily participate in the study to accept randomization for either treatment arm.
5. Signing of the approved Free and Informed Consent Form (ICF) by the Research Ethics Committee (CEP) and CONEP

Exclusion Criteria:

1. Age below 18 years
2. Patients who do not want or can fulfill the necessary home isolation for at least 14 days
3. Chronic clinical conditions, severe or not compensated, such as: insulin-dependent diabetes (types 1 or 2); uncontrolled hypertension, lung disease such as asthma or COPD; hematological and liver diseases, chronic kidney disease in advanced stage (grades 3, 4 and 5), metabolic disorders and immunosuppression
4. Use of any medication with potential interaction with CBD (such as chloroquine, clobazan, warfarin, or valproic acid) or history of undesirable reactions prior to the use of this cannabinoid
5. Inability to use oral medication
6. Pregnancy or lactation
7. History of alcohol or drug addiction
8. Smoking in the last three years
9. Marijuana use in the last three months
10. Inability to cooperate with researchers due to cognitive impairment or mental state
11. Patients with severe forms of SARS-CoV-2, (on screening, inclusion or initial visit)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-11-16 (Estimated); Study Completion 2021-11-16 (Estimated)

PRIMARY OUTCOMES:
Prevention of severe/critical stage of Covid19 | Up to 28 days
  Deterioration in clinical status from mild/moderate to severe/critical over time during the study period
Time to CoVid19 symptoms relief and number of participants with negative Clinical CoVid19 symptoms as assessed by CTCAE v5.0 | Up to 28 days
  Clinical CoVid19 symptoms Clinical improvement

SECONDARY OUTCOMES:
Change in proinflammatory cytokine concentration | Up to 28 days
  Immune reaction
Describe the parenchymal lung damage induced by COVID-19 through a qualitative analysis with chest CT | 14 days
  A qualitative CT analysis of parenchymal lung damage induced by COVID-19
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to 28 days
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Time to clinical improvement with CTCAE v5.0 CoVid19 symptoms to 0 | Up to 28 days
  Time to clinical improvement
Number of participants that need hospitalisation | Up to 28 days
  CoVid severity worsening
28-day mortality | Up to 28 days
  Mortality
Time to positive-to-negative saliva 2019-n-CoV RT-PCR conversion | Up to 28 days
  Time to negative saliva
Reduction in viral load | Up to 28 days
  Mean reduction in viral load (reduction of ≥1 log10) over time during the study period
Brief measure for assessing generalized anxiety disorder and depression | Through study completion, over time during the study period (day 0-28)]
  Brief measure for assessing generalized anxiety disorder (The GAD-7) and depression (PHQ-9)
Increment of odor detection sensitivity | Through study completion, over time during the study period (day 0-28)]
  Scores of the brief peanut butter olfactory test (Univ Florida)

CONTACTS AND LOCATIONS:
Overall Officials: Jose ALEXANDRE DE S CRIPPA, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (2):
- Brazil (2):
  - Serviço de Assistência Médica e Social do Pessoal do Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo
  - Unidade de Pronto Atendimento/UPA - 13 de Maio/Dr. Luis Atílio Losi Viana (UPA Covid), Ribeirão Preto, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately the following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. Depending on the level of the proposed use of data, approval by an independent review committee will be required for the identified purpose.

REFERENCES:
- [Derived] Crippa JAS, Pacheco JC, Zuardi AW, Guimaraes FS, Campos AC, Osorio FL, Loureiro SR, Dos Santos RG, Souza JDS, Ushirohira JM, Ferreira RR, Mancini Costa KC, Scomparin DS, Scarante FF, Pires-Dos-Santos I, Mechoulam R, Kapczinski F, Fonseca BAL, Esposito DLA, Passos ADC, Dal Fabbro AL, Bellissimo-Rodrigues F, Arruda E, Scarpelini S, Andraus MH, Nather Junior JC, Wada DT, Koenigkam-Santos M, Santos AC, Busatto Filho G, Hallak JEC. Cannabidiol for COVID-19 Patients with Mild to Moderate Symptoms (CANDIDATE Study): A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Cannabis Cannabinoid Res. 2022 Oct;7(5):658-669. doi: 10.1089/can.2021.0093. Epub 2021 Oct 7. PMID 34619044